CLINICAL TRIAL: NCT04422678
Title: Imatinib for the Treatment of SARS-COV-2 Induced Pneumonia: A Pilot Study
Brief Title: The Safety & Efficacy of Imatinib for the Treatment of SARS-COV-2 Induced Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Collaborators: Science, Technology & Innovation Funding Authority (STIFA), Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alex CCM 2020/5
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Pneumonia; ARDS; Cytokine Storm
MeSH Terms: conditions — COVID-19; Pneumonia; Cytokine Release Syndrome | interventions — Imatinib Mesylate; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Imatinib Standard Dose (Experimental): Imatinib 400 mg oral tablet once daily for 21 days
  In addition for the treatment for COVID-19 pneumonia according to the Egyptian National Protocol by the Ministry of Health (MOH).
  Interventions: Drug: Imatinib Mesylate
- Imatinib Low Dose (Experimental): Imatinib 200 mg oral tablet once daily for 21 days.
  In addition to the treatment for COVID-19 Pneumonia according to the Egyptian National Protocol by the Ministry of Health (MOH).
  Interventions: Drug: Imatinib Mesylate
- Control (Active Comparator): Treatment for COVID-19 pneumonia according to the Egyptian National Protocol by the Ministry of Health (MOH).
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Imatinib Mesylate — Adding treatment by imatinib oral tablet into the standard treatment for moderate to severe COVID-19 pneumonia.
  Other Names: Imatinib
  Arms: Imatinib Low Dose; Imatinib Standard Dose
Drug: Standard of Care — Standard of Care for the Moderate to Severe COVID-19 Pneumonia as per the Egyptian National Protocol by the Ministry of Health.
  Other Names: Standard
  Arms: Control

SUMMARY:
A randomized controlled pilot study on the safety & efficacy of imatinib for the treatment of patient with moderate to severe SARS-COV-2 induced pneumonia.

DETAILED DESCRIPTION:
As the coronavirus disease (COVID-19) spreads worldwide, awaiting the development of a vaccine, researchers are looking among the arsenal of available drugs, for a potential cure or medication to improve patients' outcome. A highly elevated levels of cytokines in COVID-19 patients requiring ICU admission, has suggested that a "cytokine storm" was associated with disease severity. Data from cellular, animal models and clinical trials, showed a beneficial role of tyrosine kinase inhibitors in the regulation of inflammation, the maintenance of endothelial barrier integrity, as well as the expression of antiviral properties. This data is especially derived from imatinib, the most studied Abl family kinase inhibitor, that is currently in clinical use for multiple medical conditions. Based on this encouraging data, we hypothesize that imatinib might be beneficial for the treatment of patients with SARS-CoV-2 pneumonia, in the aim of preventing disease progression into the severe phenotype of hypoxic respiratory failure and acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCR positive for SARS-COV-2
* Hospitalized with moderate to severe respiratory symptoms as assessed by the Egyptian Ministry of Health National Guidelines
* Informed consent explained & signed by patient or his 1st degree relatives or legally authorized representative.

Exclusion Criteria:

* Pregnant women (or) breast feeding women
* Patients younger than 18 years of age
* Patients with known allergy to imatinib
* Total bilirubin, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) > 5x upper limit of normal (ULN).
* Creatinine clearance (CrCl) < 30 mL/minute.
* Patient already on mechanical ventilation at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Disease Progression | 30 Days
  Proportion of patients with COVID-19 pneumonia progressed to critical illness in need for invasive mechanical ventilation.

SECONDARY OUTCOMES:
Improvement in Hypoxic Index | From inclusion to 30 days follow up
  Improvement of Hypoxic index( PaO2 / FiO2) calculated daily
Hospital Length of Stay | From inclusion to 30 days follow up
  Hospital Length of stay
Days on invasive mechanical ventilation | From inclusion to 30 days follow up
  Days on mechanical ventilation for patients needing intubation & invasive mechanical ventilation
Inflammatory Markers | From inclusion to 30 days
  Difference in the median levels of serum IL-6, serum ferritin, CRP at the end of the follow up period between all groups
Viral clearance | From inclusion to 30 days
  Rate of viral clearance as monitored by SARS-COV-2 PCR
Radiological assessment | From inclusion to 30 days
  Difference in the overall evaluation of pulmonary infiltrative (improving / deteriorating) as assessed by imaging (Chest X-ray or Non-contrast pulmonary CT)
Safety of Imatinib | From inclusion to 60 days
  Rate of serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Hany ASSAAD, MD, PhD, Principal Investigator — University of Alexandria

IPD SHARING:
Plan to Share IPD: No